CLINICAL TRIAL: NCT02053233
Title: Clinical Trial of Robot-assisted Training for Motor and Gait Recovery in Patients With Stroke
Brief Title: Robot-assisted Training for Stroke Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNUYH-03-2013-011
Record Dates: First submitted 2014-01-21; First posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Stroke
Keywords: stroke; robot-assisted therapy; conventional therapy; motor function
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walkbot group (Experimental): The Walkbot group received conventional physical therapy (session I for 40 min/day) companied with Walkbot training (session II for 30 min/day) 5 days a week for 4 weeks, 40 session in all. After 4-week intervention all subjects received conventional physical therapy only, 40 min/day, 5 days/week for 4 weeks.
  Interventions: Device: Walkbot group
- control group (Placebo Comparator): The control group received conventional functional rehabilitation for 40 min/session, 2 sessions/day, 5 days/week for 4 weeks, 40 sessions in all. After 4-week intervention all subjects received conventional physical therapy only, 40 min/day, 5 days/week for 4 weeks. During the test period, general rehabilitation and drug treatment can be done at the same time.
  Interventions: Device: Control group

INTERVENTIONS:
Device: Walkbot group — The physiotherapist typed patient's information then Walkbot would adjust itself to this data and the exoskeleton legs lengthen or shorten to the patient. The computer screen would provide information about speed, duration, cadence and distance. The monitor in front of the patient can offer image and feedback during the therapy process for patients.
  The whole Walkbot training process was observed by one physiotherapist and should be always ready to adjust the unloading, duration, speed and guidance force of Walkbot according to patients' different situation such as muscle spasticity, gait quality, labor-consuming and observe the changes of patients' state.
  Other Names: Walkbot
  Arms: Walkbot group
Device: Control group — The control group received conventional functional rehabilitation for 40 min/session, 2 sessions/day, 5 days/week for 4 weeks, 40 sessions in all. After 4-week intervention all subjects received conventional physical therapy only, 40 min/day, 5 days/week for 4 weeks. During the test period, general rehabilitation and drug treatment can be done at the same time.
  Other Names: conventional treatment
  Arms: control group

SUMMARY:
The robot assisted therapy is one of the new developed technologies for recovery after stroke. This study aimed to evaluating the effect of robotic gait therapy for motor recovery after stroke.

DETAILED DESCRIPTION:
This study designed an assessor-blinded, randomized, controlled clinical study. The participations followed the study protocol and were randomly divided into the control group and Walkbot group. The control group received conventional functional rehabilitation for 40 min/session, 2 sessions/day, 5 days/week for 4 weeks, 40 sessions in all. Whereas the Walkbot group received conventional physical therapy (session I for 40 min/day) companied with Walkbot training (session II for 30 min/day) 5 days a week for 4 weeks, 40 session in all. After 4-week intervention all subjects received conventional physical therapy only, 40 min/day, 5 days/week for 4 weeks. During the test period, general rehabilitation and drug treatment can be done at the same time.

ELIGIBILITY:
Inclusion Criteria:

* The subjects (age>19) with stroke 4 weeks after the onset but within 12 months were included.

Exclusion Criteria:

* Participated in the clinical studies, or received the rehabilitation therapy or therapy associated with the rehabilitation for the purpose of motor function improvement within thirty days before the start of this study.
* Cognitive disabilities or serious psychiatric illness.
* Difficulty in walking due to orthopedic problems.
* Ejection fraction less than 30% due to severe heart disease or with a diagnosis of unstable angina.
* Weight more than 135 kg or height less than 150 cm.
* Pregnancy subjects.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
function ambulation category (FAC) | within 4 weeks after robot training
  Function ambulation category was used for evaluating gait function. The outcome variable were measured immediately before treatment start (pre-training), 4 weeks after treatment (post-training) and 4 weeks after robot-treatment (follow-up). All the evaluations were done by the same professional therapist who was blind to the two group assignment.

SECONDARY OUTCOMES:
Berg balance scale (BBS) | within 4 weeks after robot training
  Berg balance scale (BBS) were used for evaluating functional performance level after training. The outcome variables were measured immediately before treatment start (pre-training), 4 weeks after treatment (post-training) and 4 weeks after robot-treatment (follow-up). All the evaluations were done by the same professional therapist who was blind to the two group assignment.
Korean modified Barthel index (K-MBI) | within 4 weeks after robot training
  Korean modified Barthel index (K-MBI) were used for evaluating functional performance level after training. The outcome variables were measured immediately before treatment start (pre-training), 4 weeks after treatment (post-training) and 4 weeks after robot-treatment (follow-up). All the evaluations were done by the same professional therapist who was blind to the two group assignment.

OTHER OUTCOMES:
EuroQol-5 dimension (EQ-5D) | within 4 weeks after robot training
  EuroQol-5 dimension (EQ-5D) was used for evaluating the effect of robot training to quality of life. The outcome variable was measured immediately before treatment start (pre-training), 4 weeks after treatment (post-training) and 4 weeks after robot-treatment (follow-up). All the evaluations were done by the same professional therapist who was blind to the two group assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Il Shin, Ph.D., Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea